CLINICAL TRIAL: NCT00588354
Title: Pilot Study of Transforaminal Epidural Injection of Clonidine for the Treatment of Acute Lumbosacral Radiculopathy
Brief Title: Epidural Clonidine for Lumbosacral Radiculopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Targeted enrollment was not reached.
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Marc A. Huntoon, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-002738; 1UL1RR024150-01 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Lumbar and Other Intervertebral Disc Disorders With Radiculopathy
Keywords: herniated disk; radiculopathy; clonidine; epidural; steroid; corticosteroid; nucleus pulposus; transforaminal
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy | interventions — Clonidine; triamcinolone hexacetonide; Triamcinolone; Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine (Experimental): Transforaminal epidural clonidine injection
  Interventions: Drug: Clonidine; Drug: Lidocaine HCl
- Steroid (Active Comparator): Transforaminal epidural steroid injection
  Interventions: Drug: Triamcinolone hexacetonide; Drug: Lidocaine HCl

INTERVENTIONS:
Drug: Clonidine — 200 or 400 micrograms clonidine
  Other Names: Catapres; Kapvay; Nexiclon
  Arms: Clonidine
Drug: Triamcinolone hexacetonide — 40 or 80 milligrams triamcinolone
  Other Names: Aristocort; Kenacort; Tri-Nasal; Triaderm; Azmacort; Trilone; Volon A; Tristoject; Tricortone
  Arms: Steroid
Drug: Lidocaine HCl — 1 ml 2% lidocaine (20 mg/mL)
  Other Names: Xylocaine; lignocaine

SUMMARY:
This was a randomized, blinded study of transforaminal epidural injection of clonidine versus a similar injection of corticosteroid for acute lumbosacral radiculopathy. The hypothesis was that clonidine will be as effective as steroid for this condition.

DETAILED DESCRIPTION:
Patients with approximately 3 months of low back pain and leg pain due to intervertebral disc herniation were randomized to transforaminal epidural injections of 2% lidocaine and either clonidine (200 or 400 micrograms) or triamcinolone (40 mg) (corticosteroid). Patients received one to three injections administered at about 2 weeks apart. Patients, investigators, and study coordinators were blinded to the treatment. The primary outcome was an 11-point Pain Intensity Numerical Rating Scale at 1 month. The hypothesis was that clonidine will be as effective as steroid for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Residents 18 years or older of Olmsted or contiguous counties and identified as having an acute unilateral radicular syndrome of less than 3 months duration (leg pain>back, discogenic cause, one or more of the following:

  * Positive Straight Leg Raise (SLR) test
  * Myotomal weakness
  * Dermatomal sensory loss) and with concordant
  * Confirmatory findings on recent MRI or CT myelogram

Exclusion Criteria:

* History of recent spinal trauma
* Cauda equina syndrome (This is a serious neurologic condition in which there is acute loss of function of the lumbar plexus, neurologic elements of the spinal canal below the termination of the spinal cord.)
* Progressive neurological deficit
* Motor deficit
* Pathological or infectious etiology
* Involvement in workers' compensation claim
* History of adverse reaction to corticosteroids, local anesthetic or clonidine
* History of one or more corticosteroid injection(s) (equivalent to 40 mg of triamcinolone acetate) in the preceding 4 months
* Pregnant
* Severe medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Huntoon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Burgher AH, Hoelzer BC, Schroeder DR, Wilson GA, Huntoon MA. Transforaminal epidural clonidine versus corticosteroid for acute lumbosacral radiculopathy due to intervertebral disc herniation. Spine (Phila Pa 1976). 2011 Mar 1;36(5):E293-300. doi: 10.1097/BRS.0b013e3181ddd597. PMID 21192304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 33 patients screened and randomized, 26 enrolled.
Pre-assignment Details: Target enrollment was not reached
Groups:
- 2% Lidocaine and Clonidine (200 or 400 ug); 2% Lidocaine and Triamcinolone (40 mg).: Patients received one to three injections administered at about 2 weeks apart. Patients,investigators, and study coordinators were blinded to the treatment.
  The primary outcome was an 11-point Pain Intensity Numerical Rating Scale at 1 month. Other outcomes included Patient Global Impression of Change and functional measures.
Period: Baseline to 2 Weeks
Arm/Group | 2% Lidocaine and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg).
Started | 11 | 15
Completed | 9 | 15
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Period: Baseline to 4 Weeks
Arm/Group | 2% Lidocaine and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg).
Started | 9 | 15
Completed | 9 | 14
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Lidocaine and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg). | Total
Number analyzed (Participants) | 11 | 15 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.4) | 50.3 (11.0) | 47.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 15 | 26
Pain Intensity Score [Mean (Standard Deviation); unit: Units on a scale] — Pain Intensity Score as measured by Pain Intensity Numerical Rating Scale (PI-NRS). This is an 11-point ordinal scale measuring patient pain, ranging from 0 (no pain) to 10 (most severe/disabling pain).
  Units on a scale | 7.0 (1.9) | 7.0 (2.0) | 7.0 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score at 4 Weeks as Measured by Pain Intensity Numerical Rating Scale (PI-NRS)
Description: 11-point ordinal scale measuring patient pain, ranging from 0 (no pain) to 10 (most severe/disabling pain).
Time Frame: 4 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 2% Lidociane and Clonidine (200 or 400 ug): Transforaminal epidural clonidine injection
- 2% Lidocaine and Triamcinolone (40 mg): Transforaminal epidural steroid injection
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 14
Units on a scale | 4.1 (2.9) | 2.7 (2.2)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.159, ANCOVA; Mean Difference (Net) = 1.54, 95% CI 2-sided [-0.52 to 3.60], Standard Error of Mean 1.05

2. Secondary Outcome: Pain Intensity Score at 2 Weeks as Measured by Pain Intensity Numerical Rating Scale (PI-NRS)
Description: 11-point ordinal scale measuring patient pain, ranging from 0 (no pain) to 10 (most severe/disabling pain).
Time Frame: 2 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 15
Units on a scale | 4.1 (2.3) | 4.0 (2.5)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.910, ANCOVA; Mean Difference (Net) = 0.11, 95% CI 2-sided [-1.79 to 2.01], Standard Error of Mean 0.97

3. Secondary Outcome: Pain Disability Score at 2 Weeks as Measured by the Roland-Morris Disability Questionnaire
Description: This scale measures functional disability due to back pain. The score of the scale is the total number of items checked, from a minimum of 0 (no disability) to a maximum of 24 (great disability). Roland MO, Morris RW. A study of the natural history of back Pain. Part 1: development of a reliable and sensitive measure of disability in low back pain. Spine 1983; 8:141-144.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 15
Units on a scale | 9.6 (5.0) | 5.7 (4.7)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.162, ANCOVA; Mean Difference (Net) = 2.96, 95% CI 2-sided [-1.04 to 6.96], Standard Error of Mean 2.04

4. Secondary Outcome: Pain Disability Score at 4 Weeks as Measured by the Roland-Morris Disability Questionnaire
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 14
Units on a scale | 9.4 (6.4) | 3.5 (4.1)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.022, ANCOVA; Mean Difference (Net) = 5.67, 95% CI 2-sided [1.22 to 10.12], Standard Error of Mean 2.27

5. Secondary Outcome: Pain Disability Score at 2 Weeks as Measured by Oswestry Low Back Pain Disability Questionnaire (ODI)
Description: This questionnaire measures a patient's permanent functional disability. The questionnaire consists of 10 sections with 6 statements each of increasing point value (from 0 to 5). The score is a percentage of the total, with higher score showing greater disability. Minimum detectable change is 10%, with a 90% CI. Change of less than this may be attributable to error in measurement.
Time Frame: 2 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 2% Lidocaine and Clonidine (200 or 400 ug): Transforaminal epidural clonidine injection
Arm/Group | 2% Lidocaine and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 15
Units on a scale | 27.0 (5.8) | 21.3 (8.4)
Statistical Analysis 1: Comparison: 2% Lidocaine and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.089, ANCOVA; Median Difference (Net) = 5.86, 95% CI 2-sided [-0.57 to 12.29], Standard Error of Mean 3.28

6. Secondary Outcome: Pain Disability Score at 4 Weeks as Measured by Oswestry Low Back Pain Disability Questionnaire
Description: as for outcome 5
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 14
Units on a scale | 23.9 (8.3) | 17.0 (6.5)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.038, ANCOVA; Mean Difference (Net) = 7.04, 95% CI 2-sided [0.83 to 13.25], Standard Error of Mean 3.17

7. Secondary Outcome: Pain Score at 2 Weeks as Measured by the Multidimensional Pain Inventory (MPI)
Description: The MPI is a comprehensive instrument comprised of 12 scales divided into three parts for assessing a number of dimensions of the chronic pain experience including pain intensity, emotional distress, cognitive and functional adaptation, and social support. Reference: Kearns RO, Turk DC, Rudy TC. The West Haven-Yale Multidimensional Pain Inventory (WHYMPI). Pain 1985; 23:345-356. Subscales were not used; the DOS WHYMPI computer program version 2.1 was used to score the instrument. Scores range from 0 (no pain) to 100 (highest pain). A score of 50 is the mean for patients with chronic pain.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 15
Units on a scale | 51.6 (10.2) | 56.0 (7.2)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.186, ANCOVA; Mean Difference (Net) = -4.83, 95% CI 2-sided [-11.75 to 2.09], Standard Error of Mean 3.53

8. Secondary Outcome: Pain Score at 4 Weeks as Measured by the Multidimensional Pain Inventory (MPI)
Description: as for outcome 7
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2% Lidociane and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg)
Number analyzed (Participants) | 9 | 14
Units on a scale | 56.7 (6.8) | 56.9 (8.2)
Statistical Analysis 1: Comparison: 2% Lidociane and Clonidine (200 or 400 ug) vs 2% Lidocaine and Triamcinolone (40 mg); Data were analyzed using analysis of covariance (ANCOVA) with baseline value included as a covariate; Test type: Superiority or Other; p = 0.918, ANCOVA; Mean Difference (Net) = -0.35, 95% CI 2-sided [-6.96 to 6.26], Standard Error of Mean 3.37

ADVERSE EVENTS:
Arm/Group | 2% Lidocaine and Clonidine (200 or 400 ug) | 2% Lidocaine and Triamcinolone (40 mg).
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 9/11 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% Lidocaine and Clonidine (200 or 400 ug) (N=11) | 2% Lidocaine and Triamcinolone (40 mg). (N=15)
Worsening of Symptoms (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Discomfort at Injection Site (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Lightheadedness (Nervous system disorders) | 5 (5) | 1 (1)
Drowsiness (Nervous system disorders) | 2 (2) | 3 (3)
Weakness (Nervous system disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; did not measure analgesia during the expected analgesic peak of bolus administration, but 10 days after last injection; compared clonidine with an active control, rather than placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No